CLINICAL TRIAL: NCT05821829
Title: Endovascular Treatment of Primary Common FEmoral Artery atheroSclerotic Disease wiTh IntraVAscular Litothripsy: the FESTIVAL Registry
Brief Title: Endovascular Treatment of Primary Common FEmoral Artery atheroSclerotic Disease wiTh IntraVAscular Litothripsy
Acronym: FESTIVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Nicola Troisi, Associate Professor of Vascular Surgery, University of Pisa
Other Study IDs: FESTIVAL
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease; Common Femoral Artery Stenosis; Common Femoral Artery Occlusion; Critical Limb-Threatening Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intravascular litothripsy (IVL) — endovascular treatment of primary common femoral artery atherosclerotic disease with intravascular litothripsy

SUMMARY:
Prospective, nonrandomized, multicenter, national, multidisciplinary, real-world data collection with the aim to evaluate the short-term safety and efficacy of intravascular lithotripsy in the treatment of steno-obstructive disease of the common femoral artery

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral arterial disease (Rutherford class 3-6)
2. Presence of a steno-obstructive lesion of the common femoral artery (Azema classification 1-3)
3. Possible endovascular treatment of both the iliac axis and/or femoro-distal vessels
4. Possible post-dilatation with plain or drug-coated balloon angioplasty

Exclusion Criteria:

1. Concomitant open surgery (ilio-femoral or femoro-distal bypass)
2. Presence of a steno-obstructive lesion of the common femoral artery in previous open surgery (Azema classification 4)
3. Presence of a steno-obstructive lesion of the common femoral artery after a previous endovascular procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severely symptomatic peripheral arterial disease and concomitant atherosclerotic de novo lesions of the common femoral artery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | Intraprocedural
  insertion/use of the device after crossing the steno-obstructive lesion and its removal without complications, restoration of vessel patency in the absence of stenosis/acute recoil >30%, rupture/perforation of the common femoral artery, need for a bailout stenting
Clinical success | Intraprocedural / 1 month
  absence of intraprocedural complications including distal embolization and improvement of at least 1 Rutherford class assessed 1 month after the procedure
Primary patency | 1 month / 6 months / 1 year
  patency of the treated vessel in the absence of a restenosis >30%
Primary assisted patency | 1 month / 6 months / 1 year
  patency of the treated vessel after one or more endovascular reinterventions
Secondary patency | 1 month / 6 months / 1 year
  patency of the treated vessel after occlusione and treatment by surgical or endovascular means
Clinically driven freedom from target lesion restenosis (cdTLR) | 1 month / 6 months / 1 year
  restenosis resulting in vessel occlusion or stenosis with maximum PSV > 2.5 m/sec

SECONDARY OUTCOMES:
Freedom from any reinterventions | 1 month / 6 months / 1 year
Patency of profunda femoris | 1 month / 6 months / 1 year
Limb salvage | 1 month / 6 months / 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

REFERENCES:
- [Result] Baig M, Kwok M, Aldairi A, Imran HM, Khan MS, Moustafa A, Hyder ON, Saad M, Aronow HD, Soukas PA. Endovascular Intravascular Lithotripsy in the Treatment of Calcific Common Femoral Artery Disease: A Case Series With an 18-Month Follow-Up. Cardiovasc Revasc Med. 2022 Oct;43:80-84. doi: 10.1016/j.carrev.2022.05.003. Epub 2022 May 7. PMID 35595607
- [Result] Wong CP, Chan LP, Au DM, Chan HWC, Chan YC. Efficacy and Safety of Intravascular Lithotripsy in Lower Extremity Peripheral Artery Disease: A Systematic Review and Meta-Analysis. Eur J Vasc Endovasc Surg. 2022 Mar;63(3):446-456. doi: 10.1016/j.ejvs.2021.10.035. Epub 2021 Dec 6. PMID 34887206
- [Result] Tepe G, Brodmann M, Werner M, Bachinsky W, Holden A, Zeller T, Mangalmurti S, Nolte-Ernsting C, Bertolet B, Scheinert D, Gray WA; Disrupt PAD III Investigators. Intravascular Lithotripsy for Peripheral Artery Calcification: 30-Day Outcomes From the Randomized Disrupt PAD III Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1352-1361. doi: 10.1016/j.jcin.2021.04.010. PMID 34167675